CLINICAL TRIAL: NCT01790334
Title: Comparing the Size of the Vena Jugular Interna Under Spontaneous Ventilation and Different Mechanical Ventilation Modes When Head is in Neutral and 30 Degree Lateral Position:Clinical Trial
Brief Title: Effects of Different Modes of Ventilation and Head Position on Size of Vena Jugular Interna
Acronym: USG-IJV
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assoc.Prof. M.D., Istanbul University
Other Study IDs: 32488
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-02

CONDITIONS: Central Line Complication
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Spontenous Ventilation (Group S): ultrasonography of Right internal jugular vein
  Interventions: Other: Ultrasonography
- Pressure control Ventilation (Group P): ultrasonography of Right internal jugular vein
  Interventions: Other: Ultrasonography
- Volume control ventilation (Group V): ultrasonography of Right internal jugular vein
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography
  Other Names: The crosssectional area and diameter of right internal jugular vein will be measured by ultrasonography

SUMMARY:
It is widely known that positive mechanical ventilation increases the positive intrathoracic pressure which affects the pressure in the RIJV, resulting in an increase of the CSA. Currently, there appears to be a lack of studies in the literature that assess the effects of different modes of ventilation of this increase.

The aim of our study is to evaluate the changes in cross-sectional area and diameters of RIJV under two different mechanical ventilation modes (PCV and VCV) and spontaneous ventilation in head neutral and 30 degree rotated lateral position by using ultrasonography and to determine the ventilation mode that is most suitable for catheterization.

ELIGIBILITY:
Inclusion Criteria:

* 30 ASA status I-II patients between 18-80 years old undergoing elective abdominal surgery

Exclusion Criteria:

* Patients with a history of congestive heart failure, pulmonary hypertension, chronic renal failure, diabetes mellitus, rheumatological diseases, neck surgery, valvular disease, obesity or RIJV catheterization will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 ASA status I-II patients between 18-80 years old undergoing elective abdominal surgery under endotracheal intubation will be included in this random, prospective, clinical study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
comparing the size of right internal jugular vein in different mechanical ventilation modes | 1 month

SECONDARY OUTCOMES:
effect of different head positions on the right internal jugular vein size | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Result] Lobato EB, Florete OG Jr, Paige GB, Morey TE. Cross-sectional area and intravascular pressure of the right internal jugular vein during anesthesia: effects of Trendelenburg position, positive intrathoracic pressure, and hepatic compression. J Clin Anesth. 1998 Feb;10(1):1-5. doi: 10.1016/s0952-8180(97)00189-x. PMID 9526929